CLINICAL TRIAL: NCT05859061
Title: Intraoperative Cryoanalgesia for Pain Management After Sternotomy: A Randomized Pilot Trial
Brief Title: Cryoanalgesia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sawyer Naze, Assistant Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00218457
Record Dates: First submitted 2023-04-13; First posted 2023-05-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoanalgesia (Experimental): Intraoperative analgesic administration will be at the discretion of the anesthesia provider. Once adequate hemostasis is achieved and prior to sternal wire placement and chest closure, patients will undergo cryoablation of bilateral T2 - T6 intercostal nerves. The cryoprobe will be positioned under direct visualization and ablation of the intercostal nerve will be performed 2-4 cm lateral to the internal mammary artery near the mid-clavicular line. Each cryoablation at -50°C to -70°C will be applied for 120 seconds to sustain an ablation length of 2-3 cm at each intercostal nerve (bilateral T2 - T6).
  Interventions: Device: cryoICE® system (AtriCure, Inc) with CryoSphere (CryoS) probe
- Standard of Care (Control) (No Intervention): Patients in this arm will receive standard of care pain management alone.

INTERVENTIONS:
Device: cryoICE® system (AtriCure, Inc) with CryoSphere (CryoS) probe — Per manufacturer instructions, the cryoprobe will be positioned under direct visualization and ablation of the intercostal nerve will be performed 2-4 cm lateral to the internal mammary artery near the mid-clavicular line. The study team plans to perform each cryoablation (-50°C to -70°C) for 120 seconds to sustain an ablation length of 2-3 cm at each intercostal nerve (bilateral T2 - T6). The probe will be removed after defrosting to avoid mechanical damage to the intercostal nerve. Cryoablation will be performed once hemostasis is achieved and prior to sternal wire placement and chest closure by a provider from the cardiac surgery team.
  Other Names: Cryoablation
  Arms: Cryoanalgesia

SUMMARY:
This study will investigate the feasibility of cryoanalgesia in patients undergoing cardiac surgery via a median sternotomy. Cryoanalgesia is a technique that uses extremely cold temperatures to temporarily ablate nerves and block pain signals. Cryoanalgesia has been used for decades for pain control after thoracic surgery and has been associated with decreased opioid consumption, decreased pain scores, and shorter hospital stays. The results of this study may lead to a useful alternative for pain control in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective CABG (coronary artery bypass graft) or single valve surgery via median sternotomy
* Reasonable expectation to be extubated within 24 hours postop

Exclusion Criteria:

* Prior history of surgery to the thorax (sternotomy, thoracotomy, thoracoscopy)
* Hemisternotomy approach
* History of cold urticaria, cryoglobulinemia, Raynaud's disease, or diabetic neuropathy
* Preoperative use of opioids
* History of chronic pain or associated syndromes
* Concurrent Cox maze procedure
* Need for post-bypass mechanical circulatory support (ECMO, IABP) or open chest
* Women who are pregnant or breastfeeding
* Patients who are unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Average Daily Opioid Consumption in MME | 48 hours
  The average daily opioid consumption in morphine milligram equivalents (MME) during the first 48 hours postoperatively serves as the study's primary outcome.

SECONDARY OUTCOMES:
Quality of Recovery Score | 48 hours/POD2 (post-operative day 2), 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: Quality of Recovery Score Scale Values: 0 - 18 Higher score means a better outcome.
Patient Satisfaction with Pain Control Regimen | 24 hours/POD1 (post-operative day 1), 48 hours/POD2, 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: IPO (International Pain Outcomes) Questionnaire Scale Values: 0 - 320 Higher score means a worse outcome.
Pain Quality | 24 hours/POD1 (post-operative day 1), 48 hours/POD2, 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: IPO (International Pain Outcomes) Questionnaire Scale Values: 0 - 320 Higher score means a worse outcome.
Pain Quality | 24 hours/POD1 (post-operative day 1), 48 hours/POD2, 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: S-LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) Pain Score Scale Values: 0-24 Higher score means a worse outcome.
Pain Severity | 24 hours/POD1 (post-operative day 1), 48 hours/POD2, 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: S-LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) Pain Score Scale Values: 0-24 Higher score means a worse outcome.
Pain Severity | 24 hours/POD1 (post-operative day 1), 48 hours/POD2, 10 days +/- 4 days, 90 days +/- 14 days, & 180 days +/- 30 days
  Scale Title: Numeric Pain Rating Scale Scale Values: 0-10 Higher score means a worse outcome.
Average Daily Pain Scores | during the first 48 hours postoperatively (starting upon ICU arrival)
  Scale Title: CPOT (Critical-Care Pain Observation Tool) Scale Values: 0-8 Higher score means a worse outcome.
Average Daily Pain Scores | during the first 48 hours postoperatively (starting upon ICU arrival)
  Scale Title: NRS (Numeric Rating Scale) Scale Values: 0-10 Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Nachiyunde B, Lam L. The efficacy of different modes of analgesia in postoperative pain management and early mobilization in postoperative cardiac surgical patients: A systematic review. Ann Card Anaesth. 2018 Oct-Dec;21(4):363-370. doi: 10.4103/aca.ACA_186_17. PMID 30333328
- [Background] Raj N. Regional anesthesia for sternotomy and bypass-Beyond the epidural. Paediatr Anaesth. 2019 May;29(5):519-529. doi: 10.1111/pan.13626. PMID 30861264
- [Background] Kar P, Ramachandran G. Pain relief following sternotomy in conventional cardiac surgery: A review of non neuraxial regional nerve blocks. Ann Card Anaesth. 2020 Apr-Jun;23(2):200-208. doi: 10.4103/aca.ACA_241_18. PMID 32275036
- [Background] Pala AA, Urcun YS, Cicek OF, Sahin S. Can Continuous Local Anesthetic Infusion After Median Sternotomy Reduce Opioid Use? Cureus. 2020 Sep 29;12(9):e10711. doi: 10.7759/cureus.10711. PMID 33133875
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882
- [Background] Katz J, Nelson W, Forest R, Bruce DL. Cryoanalgesia for post-thoracotomy pain. Lancet. 1980 Mar 8;1(8167):512-3. doi: 10.1016/s0140-6736(80)92766-x. PMID 6102235
- [Background] Graves CE, Moyer J, Zobel MJ, Mora R, Smith D, O'Day M, Padilla BE. Intraoperative intercostal nerve cryoablation During the Nuss procedure reduces length of stay and opioid requirement: A randomized clinical trial. J Pediatr Surg. 2019 Nov;54(11):2250-2256. doi: 10.1016/j.jpedsurg.2019.02.057. Epub 2019 Mar 17. PMID 30935731
- [Background] Park R, Coomber M, Gilron I, Shanthanna H. Cryoanalgesia for postsurgical pain relief in adults: A systematic review and meta-analysis. Ann Med Surg (Lond). 2021 Aug 5;69:102689. doi: 10.1016/j.amsu.2021.102689. eCollection 2021 Sep. PMID 34408872
- [Background] Lau WC, Shannon FL, Bolling SF, Romano MA, Sakwa MP, Trescot A, Shi L, Johnson RL, Starnes VA, Grehan JF. Intercostal Cryo Nerve Block in Minimally Invasive Cardiac Surgery: The Prospective Randomized FROST Trial. Pain Ther. 2021 Dec;10(2):1579-1592. doi: 10.1007/s40122-021-00318-0. Epub 2021 Sep 20. PMID 34545530
- [Background] Rijkenberg S, Stilma W, Bosman RJ, van der Meer NJ, van der Voort PHJ. Pain Measurement in Mechanically Ventilated Patients After Cardiac Surgery: Comparison of the Behavioral Pain Scale (BPS) and the Critical-Care Pain Observation Tool (CPOT). J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1227-1234. doi: 10.1053/j.jvca.2017.03.013. Epub 2017 Mar 15. PMID 28800982
- [Background] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Background] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- [Background] Rothaug J, Zaslansky R, Schwenkglenks M, Komann M, Allvin R, Backstrom R, Brill S, Buchholz I, Engel C, Fletcher D, Fodor L, Funk P, Gerbershagen HJ, Gordon DB, Konrad C, Kopf A, Leykin Y, Pogatzki-Zahn E, Puig M, Rawal N, Taylor RS, Ullrich K, Volk T, Yahiaoui-Doktor M, Meissner W. Patients' perception of postoperative pain management: validation of the International Pain Outcomes (IPO) questionnaire. J Pain. 2013 Nov;14(11):1361-70. doi: 10.1016/j.jpain.2013.05.016. Epub 2013 Sep 7. PMID 24021577
- [Background] Bauman ZM, Loftus J, Raposo-Hadley A, Samuel S, Ernst W, Evans CH, Cemaj S, Kaye AJ. Surgical stabilization of rib fractures combined with intercostal nerve cryoablation proves to be more cost effective by reducing hospital length of stay and narcotics. Injury. 2021 May;52(5):1128-1132. doi: 10.1016/j.injury.2021.02.009. Epub 2021 Feb 6. PMID 33593526
- [Background] Salenger R, Holmes SD, Rea A, Yeh J, Knott K, Born R, Boss MJ, Barr LF. Cardiac Enhanced Recovery After Surgery: Early Outcomes in a Community Setting. Ann Thorac Surg. 2022 Jun;113(6):2008-2017. doi: 10.1016/j.athoracsur.2021.06.072. Epub 2021 Aug 2. PMID 34352198
- [Background] Myles PS. More than just morbidity and mortality - quality of recovery and long-term functional recovery after surgery. Anaesthesia. 2020 Jan;75 Suppl 1:e143-e150. doi: 10.1111/anae.14786. PMID 31903564